CLINICAL TRIAL: NCT05318612
Title: (Cost)Effectiveness of MR-guided LITT Therapy in Patients With Primary Irresectable Glioblastoma: a Prospective Multicenter Randomized Controlled Trial (EMITT)
Brief Title: Effectiveness of MR-guided LITT Therapy in Irresectable Glioblastoma (EMITT)
Acronym: EMITT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch National Health Care Institute (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL79202.091.21
Record Dates: First submitted 2022-03-23; First posted 2022-04-08 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-09

CONDITIONS: Primary Glioblastoma
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, open-label randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (biopsy group) (Other): Standard of care: biopsy + adjuvant treatment
  Interventions: Procedure: Biopsy
- Intervention group (LITT group) (Experimental): Biopsy + LITT + adjuvant treatment
  Interventions: Procedure: Laser Interstitial Thermal Therapy (LITT)

INTERVENTIONS:
Procedure: Laser Interstitial Thermal Therapy (LITT) — LITT is a minimally invasive neurosurgical procedure in which a laser catheter is placed into the tumor and warms the tumor to such an extent that tumor tissue is destroyed. LITT is performed under MR-guidance.
  Arms: Intervention group (LITT group)
Procedure: Biopsy — A sample of tissue from the tumor is obtained to confirm the diagnosis.
  Arms: Control group (biopsy group)

SUMMARY:
The aim of this study is to investigate the (cost-)effectiveness of LITT (Laser Interstitial Thermal Therapy) in primary irresectable glioblastoma. Glioblastoma are the most common malignant brain tumors and are, due to their devastating nature and the fact that these tumors occur at a relatively young age (median 59 years), responsible for up to 7% of total life years lost from cancer before the age of 70.

The current treatment of glioblastoma consists of maximal safe surgery combined with adjuvant chemoradiation therapy (CRT). However, despite this aggressive treatment, these patients still face a poor prognosis (median overall survival 14.5 - 18.5 months). In addition to that, around 30% of the patients diagnosed with a glioblastoma are not suitable for surgery. These patients miss the benefit of a resection and face an even worse prognosis (median overall survival 5.1 months).

The primary aim of this project is to investigate whether laser therapy combined with CRT improves overall survival, without compromising quality of life, in comparison with CRT alone in patients with primary irresectable glioblastoma.

DETAILED DESCRIPTION:
RATIONALE: Glioblastoma (GBM) is the most common primary brain tumor with about 1000 new patients facing this diagnosis each year in the Netherlands alone. It is also one of the most devastating malignancies and due to relatively young age at presentation (median 59 years), GBMs are responsible for up to 7% of total life years lost from cancer before the age of 70. Despite many efforts, patients with glioblastoma face a poor prognosis, with 2-year survival less than 20%. Current standard of care includes maximal safe surgical resection followed by adjuvant chemoradiation therapy (CRT). Subtotal and gross total resection have been associated with significantly longer survival (median OS: 14.5-18.5 months; RR: 0.71-0.84) 6,7, but in 30% of patients surgery is not feasible. These patients miss the benefit of surgical resection and with CRT alone have a profoundly worse survival (median 5.1 months). Laser interstitial thermal therapy (LITT) is recently growing as a minimally invasive alternative to treat brain tumors. Multiple studies have shown the application of LITT in newly diagnosed and recurrent glioblastoma, in radiotherapy and chemotherapy resistant metastases or in tumors in difficult accessible locations, with promising initial results. A recent systematic review of current phase I/II studies in patients with newly diagnosed irresectable glioblastoma who received LITT yields a mean survival of 10.2 months, i.e. twice as long as with CRT alone (5.1 months). However, there is currently no high-quality prospective evidence directly comparing LITT with standard of care, precluding any conclusions on (cost-)effectiveness. After conducting a pilot study at Radboud University Medical Center to locally confirm safety and feasibility of LITT in patients with irresectable glioblastoma, we propose a prospective multicenter randomized controlled study to evaluate (cost-)effectiveness of this technique.

OBJECTIVE: The primary objective is to prove an improvement in survival without substantially compromising quality-of-life (QoL) in patients with primary irresectable glioblastoma (GBM) treated with LITT plus chemoradiation therapy (CRT) vs. CRT alone.

STUDY DESIGN: Prospective multicenter randomized controlled trial. Study population: Adult (>18 years old) patients with a radiologically suspected diagnosis of primary glioblastoma not amenable for surgical resection.

INTERVENTION: Patients will be randomized to receive either (i) biopsy and LITT, followed by standard CRT or (ii) biopsy alone, followed by standard CRT.

MAIN STUDY PARAMETERS/ENDPOINTS: The primary endpoints are overall survival (OS) and quality-of-life (QoL) using QLQ-C30+BN20 questionnaire 5 months after randomization.

Secondary endpoints are disease-specific and progression-free survival (PFS), generic QoL using EQ5D-5L and QLQ-C30+BN20, complication rates, tumor volume response, effects on adjuvant treatment and costs.

NATURE AND EXTENT OF THE BURDER AND RISKS ASSOCIATED WITH PARTICIPATION, BENEFIT AND GROUP RELATEDNESS: We hypothesize that the addition of LITT provides patients with an irresectable glioblastoma a relevant survival benefit without compromising their quality of life as compared to current standard treatment. LITT has been shown to carry limited risk of post-operative complications, mostly reversible, and has been associated with fast recovery post-treatment. The main risks associated to the procedure are bleeding, brain edema, neurological deterioration, operation site infection, epilepsy. The results of our near-finished pilot study are showing that the procedure seems to be safe and feasible.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, age >18 years
* Suspected glioblastoma
* Supratentorial localization
* Patient is not amendable for surgical resection as decided by the tumor board
* Safe trajectory/trajectories possible for ablation of at least 70% of the tumor, avoiding eloquent structures
* Karnofsky Performance Status (KPS) >=70

Exclusion Criteria:

* Contra-indication for general anesthesia or MRI
* Non-glioblastoma diagnosis on pathology analysis
* No final pathology available
* Pregnancy
* Insufficient command of the Dutch language by the patient or a family member, making it impossible to fill in the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Depending on which event occurs first: either when a study participant dies or at the end of the trial (61 months).
  Percentage of patients still alive for a given period of time after randomization.
Health Related Quality of Life (HR-QoL) | At 5 months after randomization
  QoL measured with the QLQ-C30BN20 at 5 months after randomization.

SECONDARY OUTCOMES:
Costs | At 1, 2, 3, 4, 5, 6, 12, 18, 30, 42 and 54 months after randomization.
  Use of care and health-related costs measured using costs questionnaires.
Ablation rate | Using the MRI made right after LITT procedure
  Measuring the expected ablation rate.
Progression Free Survival (PFS) | During the entire study period, estimated 18 months for each patient
  The length of time during and after the treatment of the disease that a patient lives with the disease but it does not get worse.
Disease Specific Survival (DSS) | During the entire study period, estimated 18 months for each patient
  The percentage of patients who have not died from glioblastoma.
Complication rate | During the entire study period, estimated 18 months for each patient
  Registration of complications in both study groups.
Overall survival since intervention | During the entire study period, estimated 18 months for each patient
  Percentage of patients still alive for a given period of time after surgery.
Tumor volume response | Using the MRI made right after LITT procedure
  Response of tumor tissue to LITT.
Effects of LITT on adjuvant treatment | During the entire study period, estimated 18 months for each patient
  Effects of LITT on the effect of adjuvant treatment assessed by tumor response to chemotherapy and radiotherapy on follow-up MRI.
General Quality of Life | At randomization, 72 hours after surgery, 1, 2, 3, 4, 5, 6, 12, 18, 30, 42 and 54 months after randomization.
  QoL measured with the QoL questionnaires.
Longitudinal effects | During the entire study period, estimated 18 months for each patient.
  Changes attributable to aging during the study period. Longitudinal effects will be assessed using mixed model analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mark ter Laan, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (7):
- Netherlands (7):
  - Amsterdam Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Elisabeth Tweesteden Ziekenhuis, Tilburg
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other researchers. All data will be made findable and shared for reuse and/or verification. Restrictions on data sharing only apply to MRI images due to privacy. Metadata will be published in a data repository (Radboud Data Repository). This way the data is findable. When desired, external researchers can request our data.

REFERENCES:
- [Background] Incidentie Hersentumoren. IKNL. https://www.iknl.nl/kankersoorten/hersentumoren/registratie/incidentie. Accessed October 7, 2020.
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- [Background] Rouse C, Gittleman H, Ostrom QT, Kruchko C, Barnholtz-Sloan JS. Years of potential life lost for brain and CNS tumors relative to other cancers in adults in the United States, 2010. Neuro Oncol. 2016 Jan;18(1):70-7. doi: 10.1093/neuonc/nov249. Epub 2015 Oct 12. PMID 26459813
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Weller M, van den Bent M, Hopkins K, Tonn JC, Stupp R, Falini A, Cohen-Jonathan-Moyal E, Frappaz D, Henriksson R, Balana C, Chinot O, Ram Z, Reifenberger G, Soffietti R, Wick W; European Association for Neuro-Oncology (EANO) Task Force on Malignant Glioma. EANO guideline for the diagnosis and treatment of anaplastic gliomas and glioblastoma. Lancet Oncol. 2014 Aug;15(9):e395-403. doi: 10.1016/S1470-2045(14)70011-7. PMID 25079102
- [Background] Brown TJ, Brennan MC, Li M, Church EW, Brandmeir NJ, Rakszawski KL, Patel AS, Rizk EB, Suki D, Sawaya R, Glantz M. Association of the Extent of Resection With Survival in Glioblastoma: A Systematic Review and Meta-analysis. JAMA Oncol. 2016 Nov 1;2(11):1460-1469. doi: 10.1001/jamaoncol.2016.1373. PMID 27310651
- [Background] De Witt Hamer PC, Ho VKY, Zwinderman AH, Ackermans L, Ardon H, Boomstra S, Bouwknegt W, van den Brink WA, Dirven CM, van der Gaag NA, van der Veer O, Idema AJS, Kloet A, Koopmans J, Ter Laan M, Verstegen MJT, Wagemakers M, Robe PAJT; Quality Registry Neuro Surgery glioblastoma working group from the Dutch Society of Neurosurgery. Between-hospital variation in mortality and survival after glioblastoma surgery in the Dutch Quality Registry for Neuro Surgery. J Neurooncol. 2019 Sep;144(2):313-323. doi: 10.1007/s11060-019-03229-5. Epub 2019 Jun 24. PMID 31236819
- [Background] Haj A, Doenitz C, Schebesch KM, Ehrensberger D, Hau P, Putnik K, Riemenschneider MJ, Wendl C, Gerken M, Pukrop T, Brawanski A, Proescholdt MA. Extent of Resection in Newly Diagnosed Glioblastoma: Impact of a Specialized Neuro-Oncology Care Center. Brain Sci. 2017 Dec 25;8(1):5. doi: 10.3390/brainsci8010005. PMID 29295569
- [Background] Ashraf O, Patel NV, Hanft S, Danish SF. Laser-Induced Thermal Therapy in Neuro-Oncology: A Review. World Neurosurg. 2018 Apr;112:166-177. doi: 10.1016/j.wneu.2018.01.123. Epub 2018 Feb 2. PMID 29410102
- [Background] Viozzi I, Guberinic A, Overduin CG, Rovers MM, Ter Laan M. Laser Interstitial Thermal Therapy in Patients with Newly Diagnosed Glioblastoma: A Systematic Review. J Clin Med. 2021 Jan 19;10(2):355. doi: 10.3390/jcm10020355. PMID 33477796
- [Background] Williams D, Loshak H. Laser Interstitial Thermal Therapy for Epilepsy and/or Brain Tumours: A Review of Clinical Effectiveness and Cost-Effectiveness [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2019 Jun 17. Available from http://www.ncbi.nlm.nih.gov/books/NBK545597/ PMID 31449372
- [Background] Weller M, van den Bent M, Preusser M, Le Rhun E, Tonn JC, Minniti G, Bendszus M, Balana C, Chinot O, Dirven L, French P, Hegi ME, Jakola AS, Platten M, Roth P, Ruda R, Short S, Smits M, Taphoorn MJB, von Deimling A, Westphal M, Soffietti R, Reifenberger G, Wick W. EANO guidelines on the diagnosis and treatment of diffuse gliomas of adulthood. Nat Rev Clin Oncol. 2021 Mar;18(3):170-186. doi: 10.1038/s41571-020-00447-z. Epub 2020 Dec 8. PMID 33293629
- [Background] Maringwa J, Quinten C, King M, Ringash J, Osoba D, Coens C, Martinelli F, Reeve BB, Gotay C, Greimel E, Flechtner H, Cleeland CS, Schmucker-Von Koch J, Weis J, Van Den Bent MJ, Stupp R, Taphoorn MJ, Bottomley A; EORTC PROBE Project and Brain Cancer Group. Minimal clinically meaningful differences for the EORTC QLQ-C30 and EORTC QLQ-BN20 scales in brain cancer patients. Ann Oncol. 2011 Sep;22(9):2107-2112. doi: 10.1093/annonc/mdq726. Epub 2011 Feb 15. PMID 21324954
- [Background] Taphoorn MJ, Stupp R, Coens C, Osoba D, Kortmann R, van den Bent MJ, Mason W, Mirimanoff RO, Baumert BG, Eisenhauer E, Forsyth P, Bottomley A; European Organisation for Research and Treatment of Cancer Brain Tumour Group; EORTC Radiotherapy Group; National Cancer Institute of Canada Clinical Trials Group. Health-related quality of life in patients with glioblastoma: a randomised controlled trial. Lancet Oncol. 2005 Dec;6(12):937-44. doi: 10.1016/S1470-2045(05)70432-0. PMID 16321761
- [Background] Garside R, Pitt M, Anderson R, Rogers G, Dyer M, Mealing S, Somerville M, Price A, Stein K. The effectiveness and cost-effectiveness of carmustine implants and temozolomide for the treatment of newly diagnosed high-grade glioma: a systematic review and economic evaluation. Health Technol Assess. 2007 Nov;11(45):iii-iv, ix-221. doi: 10.3310/hta11450. PMID 17999840
- [Background] Medvid R, Ruiz A, Komotar RJ, Jagid JR, Ivan ME, Quencer RM, Desai MB. Current Applications of MRI-Guided Laser Interstitial Thermal Therapy in the Treatment of Brain Neoplasms and Epilepsy: A Radiologic and Neurosurgical Overview. AJNR Am J Neuroradiol. 2015 Nov;36(11):1998-2006. doi: 10.3174/ajnr.A4362. Epub 2015 Jun 25. PMID 26113069
- [Background] McDannold NJ, Jolesz FA. Magnetic resonance image-guided thermal ablations. Top Magn Reson Imaging. 2000 Jun;11(3):191-202. doi: 10.1097/00002142-200006000-00005. PMID 11145211
- [Background] Leuthardt EC, Duan C, Kim MJ, Campian JL, Kim AH, Miller-Thomas MM, Shimony JS, Tran DD. Hyperthermic Laser Ablation of Recurrent Glioblastoma Leads to Temporary Disruption of the Peritumoral Blood Brain Barrier. PLoS One. 2016 Feb 24;11(2):e0148613. doi: 10.1371/journal.pone.0148613. eCollection 2016. PMID 26910903
- [Background] Mohammadi AM, Hawasli AH, Rodriguez A, Schroeder JL, Laxton AW, Elson P, Tatter SB, Barnett GH, Leuthardt EC. The role of laser interstitial thermal therapy in enhancing progression-free survival of difficult-to-access high-grade gliomas: a multicenter study. Cancer Med. 2014 Aug;3(4):971-9. doi: 10.1002/cam4.266. Epub 2014 May 9. PMID 24810945
- [Background] Ahluwalia M, Barnett GH, Deng D, Tatter SB, Laxton AW, Mohammadi AM, Leuthardt E, Chamoun R, Judy K, Asher A, Essig M, Dietrich J, Chiang VL. Laser ablation after stereotactic radiosurgery: a multicenter prospective study in patients with metastatic brain tumors and radiation necrosis. J Neurosurg. 2019 Mar 1;130(3):804-811. doi: 10.3171/2017.11.JNS171273. Epub 2018 May 4. PMID 29726782
- [Background] Rennert RC, Khan U, Bartek J, Tatter SB, Field M, Toyota B, Fecci PE, Judy K, Mohammadi AM, Landazuri P, Sloan AE, Kim AH, Leuthardt EC, Chen CC. Laser Ablation of Abnormal Neurological Tissue Using Robotic Neuroblate System (LAANTERN): Procedural Safety and Hospitalization. Neurosurgery. 2020 Apr 1;86(4):538-547. doi: 10.1093/neuros/nyz141. PMID 31076762
- [Background] Cabantog AM, Bernstein M. Complications of first craniotomy for intra-axial brain tumour. Can J Neurol Sci. 1994 Aug;21(3):213-8. doi: 10.1017/s0317167100041184. PMID 8000976
- [Background] Patel P, Patel NV, Danish SF. Intracranial MR-guided laser-induced thermal therapy: single-center experience with the Visualase thermal therapy system. J Neurosurg. 2016 Oct;125(4):853-860. doi: 10.3171/2015.7.JNS15244. Epub 2016 Jan 1. PMID 26722845
- [Background] Hawasli AH, Bagade S, Shimony JS, Miller-Thomas M, Leuthardt EC. Magnetic resonance imaging-guided focused laser interstitial thermal therapy for intracranial lesions: single-institution series. Neurosurgery. 2013 Dec;73(6):1007-17. doi: 10.1227/NEU.0000000000000144. PMID 24056317
- [Background] Stef van Buuren KG-O. mice: Multivariate Imputation by Chained Equations in R. Journal of Statistical Software 2011; Volume 45(issue 3)
- [Background] S vB. Flexible imputation of missing data, second edition: Boca Raton; 2008.
- [Background] Carreras G, Miccinesi G, Wilcock A, Preston N, Nieboer D, Deliens L, Groenvold M, Lunder U, van der Heide A, Baccini M; ACTION consortium. Missing not at random in end of life care studies: multiple imputation and sensitivity analysis on data from the ACTION study. BMC Med Res Methodol. 2021 Jan 9;21(1):13. doi: 10.1186/s12874-020-01180-y. PMID 33422019
- [Background] Kamath AA, Friedman DD, Hacker CD, Smyth MD, Limbrick DD Jr, Kim AH, Hawasli AH, Leuthardt EC. MRI-Guided Interstitial Laser Ablation for Intracranial Lesions: A Large Single-Institution Experience of 133 Cases. Stereotact Funct Neurosurg. 2017;95(6):417-428. doi: 10.1159/000485387. Epub 2018 Jan 17. PMID 29339639
- [Background] Riche M, Amelot A, Peyre M, Capelle L, Carpentier A, Mathon B. Complications after frame-based stereotactic brain biopsy: a systematic review. Neurosurg Rev. 2021 Feb;44(1):301-307. doi: 10.1007/s10143-019-01234-w. Epub 2020 Jan 4. PMID 31900737
- [Background] Jackson C, Westphal M, Quinones-Hinojosa A. Complications of glioma surgery. Handb Clin Neurol. 2016;134:201-18. doi: 10.1016/B978-0-12-802997-8.00012-8. PMID 26948356
- [Background] Rahmathulla G, Recinos PF, Kamian K, Mohammadi AM, Ahluwalia MS, Barnett GH. MRI-guided laser interstitial thermal therapy in neuro-oncology: a review of its current clinical applications. Oncology. 2014;87(2):67-82. doi: 10.1159/000362817. Epub 2014 Jul 3. PMID 24994550
- [Background] Franck P, Henderson PW, Rothaus KO. Basics of Lasers: History, Physics, and Clinical Applications. Clin Plast Surg. 2016 Jul;43(3):505-13. doi: 10.1016/j.cps.2016.03.007. PMID 27363764
- [Background] Di L, Wang CP, Shah AH, Eichberg DG, Semonche AM, Sanjurjo AD, Luther EM, Jermakowicz WJ, Komotar RJ, Ivan ME. A Cohort Study on Prognostic Factors for Laser Interstitial Thermal Therapy Success in Newly Diagnosed Glioblastoma. Neurosurgery. 2021 Aug 16;89(3):496-503. doi: 10.1093/neuros/nyab193. PMID 34156076
- [Background] Patel NV, Jethwa PR, Shetty A, Danish SF. Does the real-time thermal damage estimate allow for estimation of tumor control after MRI-guided laser-induced thermal therapy? Initial experience with recurrent intracranial ependymomas. J Neurosurg Pediatr. 2015 Apr;15(4):363-71. doi: 10.3171/2014.10.PEDS13698. Epub 2015 Jan 16. PMID 25580512
- [Background] Nakagawa M, Matsumoto K, Higashi H, Furuta T, Ohmoto T. Acute effects of interstitial hyperthermia on normal monkey brain--magnetic resonance imaging appearance and effects on blood-brain barrier. Neurol Med Chir (Tokyo). 1994 Oct;34(10):668-75. doi: 10.2176/nmc.34.668. PMID 7529367
- [Background] Rieke V, Butts Pauly K. MR thermometry. J Magn Reson Imaging. 2008 Feb;27(2):376-90. doi: 10.1002/jmri.21265. PMID 18219673
- [Derived] Neutel CLG, Viozzi I, Overduin CG, Rijpma A, Grutters JPC, Hannink G, van Eijsden P, Robe PA, Rovers MM, Ter Laan M. Study protocol for a multicenter randomised controlled trial on the (cost)effectiveness of biopsy combined with same-session MR-guided LITT versus biopsy alone in patients with primary irresectable glioblastoma (EMITT trial). BMC Cancer. 2023 Aug 23;23(1):788. doi: 10.1186/s12885-023-11282-7. PMID 37612610